CLINICAL TRIAL: NCT03863210
Title: Association of the State Hope and Decisional Conflict With the Outcomes of an Educational Intervention to Decrease Cardiovascular Risk in Women: Mixed Methods Study in Primary Health Care
Brief Title: Interventional Study to Decrease Cardiovascular Risk in Women in Primary Health Care in South Croatia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Split, School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: No. IP-2014-09-7672
Record Dates: First submitted 2019-02-28; First posted 2019-03-05 (Actual); Results first posted 2020-10-09 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2019-02

CONDITIONS: Cardiovascular Risk Factor
Keywords: cardiovascular risk; patient education; hope; decisional conflict; women

ARMS (1):
- Participants who received informations about lifestyle change (Experimental)
  Interventions: Other: 60-minute lecture titled "Change of lifestyle and nutrition habits to reduce cardiovascular risk"

INTERVENTIONS:
Other: 60-minute lecture titled "Change of lifestyle and nutrition habits to reduce cardiovascular risk" — All participants were exposed to the intervention. The intervention consisted of a 60-minute lecture titled "Change of lifestyle and nutrition habits to reduce cardiovascular risk". The lecture was delivered in family medicine offices by four specialists of family medicine individually to the groups of 6-8 participants. The lecture was verbal, harmonized among four family physicians, and contained instructions for changing nutrition habits, smoking habits and instructions for increasing physical activity. At the end of the lecture, each participant received a personally tailored decision aid, which included the list of her risk factors, assessment of the 10-year risk of fatal CVD (based on the data provided by the participants before the lecture), and instructions on what she should do in terms of changing the lifestyle habits.

SUMMARY:
Patient education in lifestyle changes has a positive effect on health in individuals with cardiovascular (CV) risk Despite current positive evidence about lifestyle and dietary change in the prevention of CVD, the recommendations are still not consistently and optimally applied to women, particularly in relation to their menopausal status. More information is needed about factors that will support effective implementation of educational interventions for decreasing CV risk. The aim of our study was to analyze the effect of an educational intervention, presented as a 60-minute lecture in primary health care setting about CV risk factors to women with different menopausal status, in relation to their decisional conflict about their treatment for CV risk and hope that their health will improve according to desired expectations.

DETAILED DESCRIPTION:
The study took place in family medicine (FM) offices from 1 March to 1 September 2014. Two FM offices were in the city of Split, the capital of the Split-Dalmatian County, one office in the neighboring Adriatic island of Brač and one in the southern Adriatic island of Korčula.

All participants reported their most recent menstrual period. To assess the impact of reproductive status, we used the categorization proposed by the "Stages of Reproductive Aging Workshop" (STRAW): 1) premenopausal (PRE) women - last period reported within 61 days before the intervention; 2) perimenopausal (PERI) women - last period reported 61-365 days before the intervention; and 3) postmenopausal (POST) women - last period reported more than 365 days before the intervention.

All participants were exposed to the intervention. The intervention consisted of a 60-minute lecture titled "Change of lifestyle and nutrition habits to reduce cardiovascular risk". The lecture was delivered in family medicine offices by four specialists of family medicine individually to the groups of 6-8 participants. The lecture was verbal, harmonized among four family physicians, and contained instructions for changing nutrition habits, smoking habits and instructions for increasing physical activity. At the end of the lecture, each participant received a personally tailored decision aid, which included the list of her risk factors, assessment of the 10-year risk of fatal CVD (based on the data provided by the participants before the lecture), and instructions on what she should do in terms of changing the lifestyle habits.

The study participants first completed the Pre-study questionnaire (Questionnaire 1), which included: a) demographic data, b) attitudes and knowledge questionnaire about CV risk factors, c) decisional conflict scale (DCS), d) integrative hope scale (IHS), and e) eating habits questionnaire (20).

Attitudes and knowledge questionnaire about CV risk factors was created according to the model of "Ottawa Decision Support Tutorial".

The DCS consist of 16 items rated in a 5-point Likert-type response format, and measures individual's uncertainty toward a course of action. There are five subscales: uncertainty, informed, values clarity, support and effective decision. The scores on the total scale and subscales are calculated as a sum of items, divided by the number of items and multiplied by 25, allowing for a score range from zero (no decisional conflict) to 100 points (extreme decisional conflict). The Croatian version of the scale was previously validated.

The IHS is 23-items scale, a self-rating instrument with items being rated on a six-point Likert scale from 1, strongly disagree, to 6, strongly agree. It provides an overall score and four dimension scores, obtained by summing up the individual item scores, with negative items being rated inversely. This produces possible overall hope scores ranging from 23 to 138 with higher scores representing higher hopefulness. The scores for the sub-dimensions vary according to the number of items. The Croatian version of the scale was previously validated. Hope to be healthy at 70 and hope to reduce CV risk was assessed by a visual analogue scale from 0 to 100.

EPAT is a simple, quick, self-administered tool using an easy scoring method for accurately assessing fat and cholesterol intake. It is a reliable and valid substitute for more time-consuming food records. EPAT also provides an efficient way to monitor eating patterns of patients over time and is arranged to provide an educational message that reinforces the consumption of recommended types and numbers of servings of low-fat foods. The questionnaire was translated into Croatian by the authors and then back translated by an independent language expert to confirm the translation validity.

Ten-year risk of fatal CVD was estimated using the ACC/AHA (American College of Cardiology/American Heart Association) guidelines, based on the following data collected from the study participants: age, gender, race, total and HDL (high-density lipoprotein) cholesterol, systolic blood pressure, data about antihypertensive therapy, diabetes mellitus and smoking status.

Immediately after the lecture, the participants filled the Post-lecture questionnaire (Questionnaire 2), which included: a) attitudes and knowledge about CV risk factors, b) decisional conflict scale (DCS) and c) integrative hope scale (IHS).

Three months after the lecture, the participants filled in the last questionnaire (Questionnaire 3), which included: a) attitudes and knowledge about CV risk factors, b) decisional conflict scale (DCS), c) integrative hope scale (HIS) and d) eating habits questionnaire (EPAT). Ten-year risk of fatal CVD was also calculated at this time point.

BMI, waist and hip circumference, systolic and diastolic blood pressure, blood cholesterol, triglycerides, physical activity and smoking status were measured at each of three time points.

Six months after the intervention, we contacted the participants for the final assessment, along with their feedback on the intervention in general and their personal opinions on further improvements in their lifestyle. This feedback was in the form of a semi-structured interview conducted by the authors, the interview included 13 structured questions and 4 open-ended questions.

We preformed the thematic analysis of the answers, grouping them into theme categories. Categorization of the answers was made by the two independent assessors. After determining the categories, each answer was marked s 1 if matching to specific category or as 0 if not. Answers were used as predictors in further analysis.

After the study, we grouped the participants into those who reduced the CV risk and those that did not. We used logistic regression for all parameter we measured to identify factors contributing to the reduction in CV risk.

Chi square test was used to compare categorical variables (presented as absolute numbers and percentages). For continuous variables, presented as means with 95% confidence intervals, we used Mann-Whitney U test. P values ≤0.05 were considered statistically significant. Logistic regression was used to describe the relationships between variables. Odds ratio for each outcome were reported with 95% confidence interval. All statistical analyses were conducted using the MedCalc statistical program (version 16.2.1 MedCalc Software, Ostend, Belgium).

ELIGIBILITY:
Inclusion Criteria:

* female sex
* age 45 to 60 years
* one or more CV risk factors [overweight or obesity, i. e. body mass index (BMI) ≥25 kg/m2, and/or central obesity - waist circumference ≥88 cm, high blood pressure (systolic blood pressure ≥140 mm Hg and/or diastolic blood pressure ≥90 mm Hg), high blood cholesterol (≥5.2 mmol/L) and active smoking]
* participants on antihypertensive therapy were also included in the study

Exclusion Criteria:

* current cardiovascular disease (CVD) (ischemic heart disease, peripheral artery disease, and stroke)
* malignant diseases
* serious systemic or mental diseases

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2014-03-01; Primary Completion 2014-09-01 (Actual); Study Completion 2015-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Slavica Jurić Petričević, Principal Investigator

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study took place in family medicine offices from 1 March to 1 September 2014. Two offices were in the city of Split, one office in the island of Brač and one in the island of Korčula.
  There were 781 women in age 45 to 60. All patients responding to the inclusion criteria listed below are called by telephone or directly contacted in FM offices.
Pre-assignment Details: There were 104 women enrolled in this study, but two women came out of the study at the beginning of the study.
Period: Overall Study
Arm/Group | Participants Who Received Informations About Lifestyle Change
Started | 104 (March 1st, 2014.)
Completed | 102 (September 1st, 2014.)
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Participants Who Received Informations About Lifestyle Change
Number analyzed (Participants) | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 102
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 52.0 [50.0 to 53.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Croatia | 102
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 27 [25 to 28]
Smoking status [Count of Participants; unit: Participants] | 44
Waist circumference [Median (Inter-Quartile Range); unit: cm] | 91 [86 to 95]
Hips circumference [Median (Inter-Quartile Range); unit: cm] | 107 [106 to 111]
Systolic blood pressure [Median (Inter-Quartile Range); unit: mmHg] | 130 [130 to 140]
Diastolic blood pressure [Median (Inter-Quartile Range); unit: mmHg] | 85 [80 to 90]
Total cholesterol [Median (Inter-Quartile Range); unit: mg/dL] | 61 [59 to 64]
HDL cholesterol [Median (Inter-Quartile Range); unit: mg/dL] | 1.5 [1.4 to 1.6]
LDL cholesterol [Median (Inter-Quartile Range); unit: mg/dL] | 4.1 [3.8 to 4.4]
Anti-hypertensive therapy [Count of Participants; unit: Participants] | 35
Triglicerydes [Median (Inter-Quartile Range); unit: mm/L] | 1.4 [1.3 to 1.4]

OUTCOME MEASURES:

1. Primary Outcome: Ten Year Risk of Cardiovascular Disease (CVD)
Description: Ten-year risk of fatal CVD was estimated using the ACC/AHA (American College of Cardiology/American Heart Association) guidelines, based on the following data collected from the study participants: age, gender, race, total and HDL (high-density lipoprotein) cholesterol, systolic blood pressure, data about antihypertensive therapy, diabetes mellitus and smoking status.
Time Frame: Change from baseline 10-year risk of CVD at 3 months
Measure: Median (95% Confidence Interval); unit: percentage of risk
Arm/Group | Participants Who Received Informations About Lifestyle Change
Number analyzed (Participants) | 102
percentage of risk | 2.9 [2.2 to 3.6]

2. Primary Outcome: Decisional Conflict (DC)
Description: DC was estimated using Decisional Conflict Scale (DCS) consist of 16 items rated in a 5-point Likert-type response format, and measures individual's uncertainty toward a course of action. There are five subscales: uncertainty, informed, values clarity, support and effective decision. The scores on the total scale and subscales are calculated as a sum of items, divided by the number of items and multiplied by 25, allowing for a score range from zero (no decisional conflict) to 100 points (extreme decisional conflict). The Croatian version of the scale was previously validated.
Time Frame: Change from baseline DC at 3 months
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Participants Who Received Informations About Lifestyle Change
Number analyzed (Participants) | 102
score on a scale | 27 [25 to 30]

3. Primary Outcome: State Hope
Description: State hope was estimated using Integrative Hope Scale (IHS), 23-items scale, a self-rating instrument with items being rated on a six-point Likert scale from 1, strongly disagree, to 6, strongly agree. It provides an overall score and four dimension scores, obtained by summing up the individual item scores, with negative items being rated inversely. This produces possible overall hope scores ranging from 23 to 138 with higher scores representing higher hopefulness. The scores for the sub-dimensions vary according to the number of items. The Croatian version of the scale was previously validated.
Time Frame: Change from baseline state hope at 3 months
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Participants Who Received Informations About Lifestyle Change
Number analyzed (Participants) | 102
score on a scale | 105 [102 to 108]

4. Secondary Outcome: Waist Circumference
Time Frame: Change from baseline waist circumference at 3 months
Measure: Median (95% Confidence Interval); unit: cm
Arm/Group | Participants Who Received Informations About Lifestyle Change
Number analyzed (Participants) | 102
cm | 89 [87 to 92]

5. Secondary Outcome: Hips Circumference
Time Frame: Change from baseline hips circumference at 3 months
Measure: Median (95% Confidence Interval); unit: cm
Arm/Group | Participants Who Received Informations About Lifestyle Change
Number analyzed (Participants) | 102
cm | 107 [105 to 110]

6. Secondary Outcome: Weight
Time Frame: Change from baseline weight at 3 months
Measure: Median (95% Confidence Interval); unit: kg
Arm/Group | Participants Who Received Informations About Lifestyle Change
Number analyzed (Participants) | 102
kg | 61 [54 to 68]

ADVERSE EVENTS:
Arm/Group | Participants Who Received Informations About Lifestyle Change
All-Cause Mortality (participants affected / at risk) | 0/102
Serious Adverse Events (participants affected / at risk) | 0/102
Other Adverse Events (participants affected / at risk) | 0/102

LIMITATIONS AND CAVEATS:
These results should be considered in view of the limitation that we could not use a control group in the setting where the intervention was delivered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No